## NCT06115408

## Evaluation of Using Dienogest and N-Acetyl Cysteine on the Volume of Uterine Leiomyoma

Faculty of Medicine
Ain Shams University
2023- 2024

Table 1: Comparison between two groups regarding demographic data of patients:

| | | Group A (Dienogest) | | | Group | B (NAC) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | (N=20) | | | | (1) | N=20) | | t* | P value |
| | Range | Mean | SD | Range | Mean | SD | | | |
| Aş | ge | 23.00-45.00 | 40.30 | 6.48 | 23.00-45.00 | 38.20 | 6.57 | 1.02 | 0.32 |
| | N | | 9, | <b>6</b> | N | % | | X <sup>2**</sup> | P value |
| Residence | Urban | 15 | 75.0% | | 14 | 70.0% | | 0.13 | 0.72 |

| | Rural | 5 | 25.0% | 6 | 30.0% | | |
|------------|-----------|----|-------|----|-------|------|------|
| | Housewife | 19 | 95.0% | 19 | 95.0% | 0.00 | 1.00 |
| Occupation | Working | 1 | 5.0% | 1 | 5.0% | FE | 1.00 |

Both groups have similar age distributions, with no significant difference (p = 0.32).

The distribution of patients based on residence and occupation is also similar between the groups (P value >0.05), indicating well-matched cohorts for demographic factors.

Table 2: Comparison between two groups regarding medical history of patients:

| | | Group A | (Dienogest) | Group | B (NAC) | | |
|---|---|---|---|---|---|---|---|
| | (N=20) | | (N | V=20) | $X^{2*}$ | P value | |
| | N | % | N | % | | | |
| Special habits | No | 20 | 100.0% | 20 | 100.0% | - | - |
| Past history of gynecologic cancer No | | 20 | 100.0% | 20 | 100.0% | - | - |
| Past history of pelvic infection | nfection No | | 100.0% | 20 | 100.0% | - | - |

| Medical history | Negative | 20 | 100.0% | 20 | 100.0% | - | - |
|------------------|----------|----|--------|----|--------|------|------|
| Surgical history | Negative | 12 | 60.0% | 7 | 35.0% | 2.51 | 0.11 |
| | Positive | 8 | 40.0% | 13 | 65.0% | 2.51 | 0.11 |

<sup>\*</sup>Chi square test

There are no significant differences between the groups in terms of special habits, history of gynecologic cancer, pelvic infection, or medical history.

A notable but non-significant trend is observed in the surgical history, where Group B has a higher percentage of positive surgical history (65% vs. 40%), though this difference is not statistically significant (p = 0.11).

Table 3: Comparison between two groups regarding Gynecological history of patients:

| | | | Group A (Dienogest) (N=20) | | D B (NAC)<br>N=20) | X <sup>2*</sup> | P value |
|---|---|---|---|---|---|---|---|
| | | N | % | N | % | | |
| Decorlegity of avala | Regular | 12 | 60.0% | 10 | 50.0% | 0.40 | 0.52 |
| Regularity of cycle Irregular | | 8 | 40.0% | 10 | 50.0% | 0.40 | 0.53 |
| Contraceptive methods No | | 8 | 40.0% | 7 | 35.0% | 2.15 | 0.67 |

| | IUD | 10 | 50.0% | 10 | 50.0% | FE | |
|---|---|---|---|---|---|---|---|
| | OCP | 2 | 10.0% | 1 | 5.0% | | |
| | Tubal ligation | 0 | 0.0% | 2 | 10.0% | | |
| Previous complications from | No | 20 | 100.0% | 20 | 100.0% | - | - |
| contraceptive method | 110 | 2 | 100.070 | 2 | 100.070 | | |

<sup>\*</sup>Chi square test (FE: Fisher Exact)

Both groups show a similar distribution in terms of cycle regularity and contraceptive methods. The use of contraceptive methods like IUDs is equally common in both groups (50%), suggesting similar baseline characteristics for contraceptive use.

Table 4: Comparison between two groups regarding obstetric history of patients:

| | | Group A (Dienogest) (N=20) | | | · | p B (NAC<br>N=20) | t* | P value | |
|---|---|---|---|---|---|---|---|---|---|
| | Range | Mean | SD | Range | Mean | SD | | | |
| Duration since la | st delivery (years) | 3.50-25.00 | 11.88 | 5.38 | 2.50-20.00 | 9.73 | 6.09 | 1.06 | 0.30 |
| | | N | % | | N | 9/ | <b>6</b> | X <sup>2**</sup> | P value |
| Gravidity | avidity 0 3 | | 15.0 | 0% | 1 | 5.0% | | 8.75 | 0.47 |

| | 1 | 2 | 10.0% | 3 | 15.0% | FE | |
|-----------|-----------|----|-------|----|-------|------------|------|
| | 2 | 5 | 25.0% | 3 | 15.0% | | |
| | 3 | 3 | 15.0% | 6 | 30.0% | | |
| | 4 | 3 | 15.0% | 2 | 10.0% | | |
| | 5 | 2 | 10.0% | 1 | 5.0% | | |
| | 6 | 1 | 5.0% | 0 | 0.0% | | |
| | 7 | 1 | 5.0% | 0 | 0.0% | | |
| | 8 | 0 | 0.0% | 3 | 15.0% | | |
| | 9 | 0 | 0.0% | 1 | 5.0% | | |
| | 0 | 3 | 15.0% | 1 | 5.0% | 1.16 | |
| Gravidity | 1-3 | 10 | 50.0% | 12 | 60.0% | 1.16<br>FE | 0.73 |
| | 4 or more | 7 | 35.0% | 7 | 35.0% | FE | |
| | 0 | 3 | 15.0% | 5 | 25.0% | | |
| | 1 | 2 | 10.0% | 2 | 10.0% | | |
| | 2 | 8 | 40.0% | 3 | 15.0% | 5.70 | |
| Parity | 3 | 4 | 20.0% | 5 | 25.0% | 5.79 | 0.47 |
| | 4 | 0 | 0.0% | 2 | 10.0% | FE | |
| | 5 | 3 | 15.0% | 2 | 10.0% | | |
| | 7 | 0 | 0.0% | 1 | 5.0% | | |
| | 0 | 3 | 15.0% | 5 | 25.0% | 5.70 | |
| Parity | 1-3 | 14 | 70.0% | 10 | 50.0% | 5.79<br>FE | 0.47 |
| | 4 or more | 3 | 15.0% | 5 | 25.0% | FE | |
| | 0 | 13 | 65.0% | 8 | 40.0% | | |
| | 1 | 4 | 20.0% | 7 | 35.0% | 0.21 | 0.02 |
| Abortions | 2 | 3 | 15.0% | 0 | 0.0% | 9.21<br>FE | 0.03 |
| | 3 | 0 | 0.0% | 4 | 20.0% | _ re | |
| | 5 | 0 | 0.0% | 1 | 5.0% | | |
| Abortions | No | 13 | 65.0% | 8 | 40.0% | 2.51 | 0.11 |

| | Yes | 7 | 35.0% | 12 | 60.0% | | |
|------------------|-----------|----|-------|----|-------|------------|------|
| | 0 | 3 | 15.0% | 5 | 25.0% | | |
| | 1 | 4 | 20.0% | 2 | 10.0% | | |
| | 2 | 5 | 25.0% | 3 | 15.0% | 5.50 | |
| Living | 3 | 6 | 30.0% | 5 | 25.0% | 5.56<br>FE | 0.56 |
| C | 4 1 | | 5.0% | 4 | 20.0% | FE_ | |
| | 5 | | 5.0% | 0 | 0.0% | | |
| | 7 | 0 | 0.0% | 1 | 5.0% | | |
| | 0 | 3 | 15.0% | 5 | 25.0% | 2.70 | |
| Living | 1-3 | 15 | 75.0% | 10 | 50.0% | 2.70 | 0.29 |
| | 4 or more | 2 | 10.0% | 5 | 25.0% | FE | |
| Mode of | NVD | 7 | 41.2% | 5 | 33.3% | 0.21 | 0.65 |
| delivery (years) | CS | 10 | 58.8% | 10 | 66.7% | 0.21 | 0.03 |

The gravidity, parity, and history of abortions are distributed similarly across both groups, with no significant differences noted.

Group A shows a slightly higher mean duration since the last delivery compared to Group B, but this difference is not statistically significant (p = 0.30).

Table 5: Comparison between two groups regarding anthropometric measures of patients:

| | Group A | (Dienoge | est) | Group | B (NAC) | | | |
|---|---|---|---|---|---|---|---|---|
| | (N=20) | | | (1) | V=20) | t* | P value | |
| | Range Mean SD | | | Range | Mean | SD | | |
| Weight (Kg) | 60.00-120.00 | 78.70 | 15.04 | 60.00-95.00 | 81.20 | 9.34 | 0.63 | 0.53 |
| Height (cm) | 158.00-173.00 164.90 4.64 | | 158.00-172.00 | 166.75 | 4.46 | 1.29 | 0.21 | |
| BMI (Kg/m <sup>2</sup> ) | 22.77-46.87 | 28.98 | 5.86 | 24.03-32.11 | 29.14 | 2.54 | 0.11 | 0.91 |

## \*Student t test

There are no significant differences in weight, height, or BMI between the two groups (P value>0.05), indicating that both groups are comparable in terms of anthropometric measures.

Table 6: Comparison between two groups regarding clinical examination of patients:

| | - | (Dienoge<br>N=20) | est) | | p B (NAC<br>N=20) | ) | t* | P value |
|---|---|---|---|---|---|---|---|---|
| | Range Mean SD | | | Range | Mean | SD | | |
| Temperature | 37.00-37.00 | 37.00 | 0.00 | 37.00-37.00 | 37.00 | .00 | - | - |
| Pulse | 65.00-85.00 | 76.90 | 6.04 | 73.00-88.00 | 80.65 | 3.95 | 2.32 | 0.03 |
| Systolic BP | 90.00-120.00 | 110.50 | 9.45 | 90.00-120.00 | 106.00 | 8.83 | 1.56 | 0.13 |

| Di | iastolic BP | 60.00-80.00 | 72.00 | 8.34 | 60.00-80.00 | 67.00 | 8.65 | 1.86 | 0.07 |
|---|---|---|---|---|---|---|---|---|---|
| | | N | 9, | <b>6</b> | N | % | | X <sup>2**</sup> | P value |
| General appearance | Normal | 20 | 100.0% | | 20 | 100.0% | | - | - |
| D - 11 | No | 19 | 95.0% | | 20 | 100.0% | | 1.03 | 1.00 |
| Pallor | Yes | 1 | 5.0% | | 0 | 0.0% | | FE | 1.00 |
| Abdominal | Free | 20 | 100 | .0% | 19 | 95. | 0% | 1.03 | |
| obstetric examination | Distended abdomen | 0 | 0.0 | )% | 1 | 5.0 | )% | FE | 1.00 |
| 1 1 | Free | 16 | 80. | 0% | 11 55.0% | | 0% | 2.60 | |
| local | Vaginal bleeding | 2 | 10. | 0% | 7 | 35.0% | | 3.69 | 0.22 |
| examination | Bulky uterus | 2 | 10. | 0% | 2 | 10. | 0% | FE | |

The only significant difference observed is in the pulse rate, with Group B having a slightly higher mean pulse rate (p = 0.03). Other clinical parameters like temperature, systolic, and diastolic blood pressure do not differ significantly between the groups (P value >0.05).

Table 7: Comparison between two groups regarding volume of leiomyoma before and after treatment (largest lesion):

| | Group A (Dienogest) | | | Group B (NAC) | | | | |
|---|---|---|---|---|---|---|---|---|
| | (N=20) | | (N=20) | | | Z* | P value | |
| | Range | Median | IQR | Range | Median | IQR | | |
| Leiomyoma volume (cm³) before | 1.43-45.24 | 15.53 | 4.31-25.01 | 1.00-108.00 | 9.00 | 4.09-14.32 | 0.52 | 0.61 |

| T 1 (3) C | 2 ( ( 7 ( 2 ( | 10.54 | 0.05.20.61 | 2 24 115 00 | 12.12 | 7740416 | 0.50 | 0.62 |
|---|---|---|---|---|---|---|---|---|
| Leiomyoma volume (cm <sup>3</sup> ) after | 2.66-76.36 | 19.54 | 8.23-32.61 | 3.24-115.90 | 13.13 | /./4-24.16 | 0.50 | 0.63 |

<sup>\*</sup>Mann Whitney U test

Median leiomyoma volume slightly increases after treatment in both groups, but the differences between the groups are not statistically significant (p > 0.05), indicating that both treatments had similar effects on leiomyoma volume.





Table 8: Comparison between two groups regarding dysmenorrhea VAS score before and after treatment:

| | Group A (Dienogest) | | | Group B (NAC) | | | | |
|---|---|---|---|---|---|---|---|---|
| | (N=20) | | (N=20) | | | t* | P value | |
| | Range | Mean | SD | Range | Mean | SD | | |
| VAS score for dysmenorrhea before | 2.00-10.00 | 7.10 | 2.88 | 5.00-10.00 | 7.30 | 1.78 | 0.26 | 0.79 |
| VAS score for dysmenorrhea after | .00-8.00 | 1.35 | 2.35 | 1.00-7.00 | 3.70 | 1.69 | 3.64 | <mark>0.001</mark> |

<sup>\*</sup>Student t test

A significant reduction in VAS scores for dysmenorrhea is observed in both groups after treatment, with Group A showing a more pronounced improvement (p = 0.001).





Table 9: Comparison between two groups regarding HMB assessment before and after treatment:

| | Group A (Dienogest) | | | Gro | .C) | | | |
|---|---|---|---|---|---|---|---|---|
| | (N=20) | | | (N=20) | | | $Z^*$ | P value |
| | Range | Median | IQR | Range | Median | IQR | | |
| HMB assessment (PBAC) before | 10.00-200.00 | 70.00 | 15.00-110.00 | 10.00-200.00 | 50.00 | 15.00-90.00 | 0.9 | 0.86 |
| HMB assessment (PBAC) after | .00-200.00 | .00 | .00-9.00 | 3.00-200.00 | 25.00 | 15.00-70.00 | 4.10 | 0.00 |

<sup>\*</sup>Mann Whitney U test

Group A shows a significant reduction in PBAC scores after treatment, indicating a better response to treatment compared to Group B (P value = 0.00).





Table 10: Comparison between two groups regarding hemoglobin level before and after treatment:

| | Group A (Dienogest) | | | Grou | p B (NAC | | | |
|---|---|---|---|---|---|---|---|---|
| | (N=20) | | (N=20) | | | t* | P value | |
| | Range | Mean | SD | Range | Mean | SD | | |
| Hemoglobin level before | 7.60-12.80 | 10.54 | 1.65 | 9.30-13.60 | 11.39 | 1.46 | 1.73 | 0.09 |
| Hemoglobin level after | 8.20-13.20 | 10.99 | 1.41 | 7.90-13.80 | 11.63 | 1.51 | 1.39 | 0.17 |

<sup>\*</sup>Student t test

While hemoglobin levels increase slightly in both groups after treatment, the differences between the groups are not statistically significant (p > 0.05).





## **Comparison of outcome measures before and after treatment:**

Table 11: Comparison between outcome measures before and after treatment in group A (Dienogest):

| | Mean | SD | t* | P value |
|-----------------------------------|--------|--------------|------|---------|
| VAS score for dysmenorrhea before | 7.10 | 2.88 | 774 | 0.00 |
| VAS score for dysmenorrhea after | 1.35 | 2.35 | 7.74 | 0.00 |
| Hemoglobin level before | 10.54 | 1.65 | 2.79 | 0.01 |
| Hemoglobin level after | 10.99 | 1.41 | 2.78 | 0.01 |
| | Median | IQR | Z** | P value |
| Leiomyoma volume (cm3) before | 15.53 | 4.31-25.01 | 2.70 | 0.01 |
| Leiomyoma volume (cm3) after | 19.54 | 8.25-32.61 | 2.78 | 0.01 |
| HMB assessment (PBAC) before | 70.00 | 15.00-110.00 | 2.00 | 0.004 |
| HMB assessment (PBAC) after | 0.00 | 0.00-8.50 | 2.88 | 0.004 |

Significant improvements are observed in VAS scores, HMB assessment, and hemoglobin levels after treatment, suggesting that Dienogest is effective. But leiomyoma volume is significantly increased after treatment.

Table 12: Comparison between outcome measures before and after treatment in group B (NAC):

| | Mean | SD | t* | P value |
|-----------------------------------|--------|-------------|------|---------|
| VAS score for dysmenorrhea before | 7.30 | 1.78 | ( 10 | 0.00 |
| VAS score for dysmenorrhea after | 3.70 | 1.69 | 6.49 | 0.00 |
| Hemoglobin level before | 11.39 | 1.46 | 1 40 | 0.10 |
| Hemoglobin level after | 11.63 | 1.51 | 1.40 | 0.18 |
| | Median | IQR | Z** | P value |
| Leiomyoma volume (cm3) before | 9.00 | 4.09-14.32 | 2.46 | 0.001 |
| Leiomyoma volume (cm3) after | 13.13 | 7.74-24.16 | 3.46 | 0.001 |
| HMB assessment (PBAC) before | 50.00 | 15.00-90.00 | 1.70 | 0.00 |
| HMB assessment (PBAC) after | 25.00 | 15.00-70.00 | 1.78 | 0.08 |

Similar to Group A, Group B also shows significant improvements in VAS scores and increase in leiomyoma volume, though the changes in hemoglobin levels and HMB assessments are less pronounced.